CLINICAL TRIAL: NCT01318772
Title: Clinical Image Evaluation for the KALARE (DREX-KL80) With New Digital Camera and Image Processor
Brief Title: Clinical Image Evaluation for the DREX-KL80 Imaging System
Status: Completed | Type: Observational
Sponsor: Toshiba America Medical Systems, Inc. (Industry)
Responsible Party: Charlemagne Chua, Manager, Regulatory Affairs, Toshiba America Medical Systems
Other Study IDs: KH-001
Record Dates: First submitted 2011-03-17; First posted 2011-03-18 (Estimated); Last update posted 2011-03-18 (Estimated); Status verified 2011-03

CONDITIONS: Obtain Diagnostic Images With the New Digital Camera and Image Processor for Evaluation.
MeSH Terms: interventions — Radiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Fluoroscopy and Angiography Procedure: Patient that have been scheduled for routine diagnostic fluoroscopy and angiography procedures by their physician.
  Interventions: Device: Radiography and Fluoroscopy Imaging System

INTERVENTIONS:
Device: Radiography and Fluoroscopy Imaging System — KALARE (DREX-KL80) is a new high resolution digital system designed for digital spot imaging, with the primary goal to address R/F and DSA clinical applications and produce images in a digital format.
  The system includes a new digital camera and a new image processor.
  Other Names: KALARE (DREX-KL80)

SUMMARY:
The purpose of this study is to acquire the clinical data required by the United States Food and Drug Administration (USFDA) for 510(k) submission, for approval of a new high resolution imaging system for fluoroscopy/radiography. It is expected that the new KALARE (DREX-KL80)high resolution imaging system will meet the design specifications. A minimum of 30 cases will be submitted for evaluation of claims for intended clinical applications.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patient 18 years and older
* Not pregnant
* Not a safety risk patient

Exclusion Criteria:

* Male and female patient under 18 years old
* Pregnant subjects
* High safety risk subjects
* Subjects and/or Legal Guardian Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female patient 18 years and older
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2010-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Collection of representative images | Estimated completion 4 weeks after start of the study
  Collect 30 to 60 represenative images to support pre-market submission.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Winkler, M.D., Principal Investigator — Stienberg Diagnostic Meidcal Imaging (SDMI)
Locations (1):
- SDMI, Las Vegas, Nevada, United States